CLINICAL TRIAL: NCT05493696
Title: Effect of Antigravity Treadmill (Alter G) Training on Gait Characteristics and Balance After Healed Adult Burns: A Randomized Controlled Trial
Brief Title: Antigravity Treadmill Training on Gait Characteristics and Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umm Al-Qura University (Other)
Responsible Party: Principal Investigator, Anwar Abdelgayed Ebid, Professor Physical Therapy, Faculty of Applied Medical Sciences, Umm Al-Qura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2022-07-30; First posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Burns
Keywords: Burn; Gait; Balance; Antigravity treadmill
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (ALG+TPTP) (Experimental): Patients received Antigravity treadmill training + Traditional physical therapy program
  Interventions: Device: Antigravity treadmill; Other: Traditional physical therapy program
- Group 2 (TPTP) (Active Comparator): Patients received a Traditional physical therapy program
  Interventions: Other: Traditional physical therapy program

INTERVENTIONS:
Device: Antigravity treadmill — Alter G training for 30-minute, 3 times/week, 75% body weight
  Other Names: Traditional physical therapy program
  Arms: Group 1 (ALG+TPTP)
Other: Traditional physical therapy program — applied 3 times/week for 12 weeks

SUMMARY:
Severe burn injuries are associated with hypermetabolic responses and increased catabolism. These generalized changes lead to a vast loss of muscle mass and cause reduced muscle strength and endurance, limited walking ability, and reduced functional mobility Recently, the antigravity treadmill or lower body positive pressure (LBPP) technology has been developed as a unique system of maintaining a participant's body weight all through treadmill training and developing low-load treadmill walking using a unique treadmill system that allows gaining the benefits of low-load treadmill walking without interrupting with locomotion dynamics

DETAILED DESCRIPTION:
Objective: This single-blind randomized controlled trial aimed to examine the effects of antigravity treadmill training on gait characteristics and balance in healed adult burned patients.

Methods: Fifty-five adult burn patients were chosen to participate in this study, their ages ranged from 18 to 35 years. They were randomly allocated to Alter G (ALG) (n=22), and control (Cont) (n=23) groups. The control group received a traditional physical therapy program (TPTP), three times per week. In contrast, the experimental group received antigravity treadmill training (30 minutes,3 times/week, speed 0.1 m/sec, 75% body weight) in addition to the traditional physical therapy program given to the control group. All study participants followed the instructions recommended for the exercise performed (three days per week) in terms of intensity, type, and duration to limit any difference between groups, as well as instructions about not exercising the rest of the week. During the study period, both groups received standard medical care. outcome measures: gait characteristics and postural stability indices were measured at the baseline (pre) and end of 12 weeks of intervention (post). The Statistical Package for the Social Sciences (SPSS) software was used for statistical analysis. The Shapiro-Wilk test was used to determine the normality of the data. The paired t-test was used to test within-group comparisons of mean changes in muscle strength, gait characteristics, and postural stability indices. The unpaired t-test was used to compare between groups. P<0.05 was chosen as the level of significance.

ELIGIBILITY:
Inclusion Criteria:

* Patients with circumferential lower limb deep second to third-degree thermal injury
* Burns extending from the lower trunk to the foot were considered
* The total body surface area (TBSA) ranges from 35 to 50%
* All patients completed the same physical therapy program during hospitalization peroid

Exclusion Criteria:

* Lower limb prosthesis
* Severe musculoskeletal disorders
* Serious cardiovascular insult
* Participation in an outside physical training program
* Fracture
* Medication that negatively impacts the study's results
* Brain injury
* Vestibular disorders
* Visual disorders
* History of epilepsy

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-28 (Actual)

PRIMARY OUTCOMES:
Change in Gait characteristics | at baseline and after 12 weeks
  Stride length (cm)
Change in Gait characteristics | At baseline and after 12 weeks
  Step length (cm)
Change in Gait characteristics | At baseline and after 12 weeks
  Velocity (cm/sec)
Change in Gait characteristics | At baseline and after 12 weeks
  Cadence (step/mint)
Change in Gait characteristics | At baseline and after 12 weeks
  Double support time (sec)
Change in Postural stability indices | At baseline and after 12 weeks
  Medio-lateral Stability Index (MLI)
Change in Postural stability indices | At baseline and after 12 weeks
  Antero-posterior Stability Index (API)
Change in Postural stability indices | At baseline and after 12 weeks
  Overall Stability Index (OSI)

CONTACTS AND LOCATIONS:
Overall Officials: Anwar Ebid, PhD, Principal Investigator — Professor Physical Therapy
Locations (1):
- Faculty of Applied Medical Sciences, Mecca, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No